CLINICAL TRIAL: NCT00623701
Title: A Multicentre, Multinational, Placebo-controlled, Double-blind, Randomized Study to Evaluate Efficacy and Safety of a Perennial, Sublingual, Specific Immunotherapy in Patients With Rhinoconjunctivitis With/Without Controlled Asthma Caused by Grass Pollen
Brief Title: Efficacy and Safety From a High-dosed Sublingual Grass Pollen Preparation
Acronym: ALLEGRA6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AL0703st; 2007-000823-16 (EudraCT Number)
Record Dates: First submitted 2008-02-19; First posted 2008-02-26 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Allergy; Rhinitis; Conjunctivitis
Keywords: sublingual grass pollen preparation; IgE-mediated Allergic Disease attributed to grass pollen
MeSH Terms: conditions — Hypersensitivity; Rhinitis; Conjunctivitis | interventions — AllerSlit forte

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): sublingual placebo preparation
  Interventions: Biological: Allerslit forte
- 2 (Experimental): Sublingual preparation, 40 micro grams Phl p 5 maintenance dose
  Interventions: Biological: Allerslit forte

INTERVENTIONS:
Biological: Allerslit forte — sublingual placebo preparation, daily
  Arms: 1
Biological: Allerslit forte — Sublingual preparation, 40 micro grams Phl p 5 maintenance dose,daily
  Arms: 2

SUMMARY:
Efficacy and Safety from a high-dosed sublingual grass pollen preparation

ELIGIBILITY:
Inclusion Criteria:

* Allergic rhinoconjunctivitis attributable to grass pollen
* Positive SPT
* Positive EAST
* Positive provocation Test

Exclusion Criteria:

* Serious chronic disease
* other perennial allergies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2008-03; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Symptom and Medication Score | Grass pollen season 2009

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Reich, Professor, Principal Investigator — not affiliated
Locations (1):
- Prof. Kristian Reich, MD, Hamburg, Germany

REFERENCES:
- See also: Leader in specific allergy research and therapy — http://www.allergopharma.de
- See also: Click here for information about this trial in the European Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/trial/2007-000823-16/DE